CLINICAL TRIAL: NCT01537042
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel-group, Polysomnography Study to Investigate Safety and Efficacy of the Rotigotine Transdermal Patch in Subjects With Restless Legs Syndrome and End-Stage Renal Disease Requiring Hemodialysis
Brief Title: A Sleep Laboratory Study to Investigate the Safety and Efficacy of the Rotigotine Skin Patch in Subjects With Restless Legs Syndrome and End-Stage Renal Disease Requiring Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB BIOSCIENCES GmbH (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP0934; 2011-003486-15 (EudraCT Number)
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Results first posted 2014-11-03 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Restless Legs Syndrome; End-Stage Renal Disease
Keywords: Rotigotine; Neupro; Restless Legs Syndrome; RLS; End-Stage Renal Disease
MeSH Terms: conditions — Restless Legs Syndrome; Kidney Failure, Chronic | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rotigotine (Experimental): Rotigotine Transdermal Patch
  1 mg/24 h, 2 mg/24 h or 3 mg/24 h once daily depending on optimal dose; maximal dose is 3 mg/24 h.
  Interventions: Drug: Rotigotine
- Placebo (Placebo Comparator): Transdermal patch matched according to patch size and appearance.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rotigotine — Transdermal patch; Dose: 1 mg/24 h, 2 mg/24 h or 3 mg/24 h once daily depending on optimal dose; maximal dose is 3 mg/24 h.
  Subjects start with a Rotigotine dose of 1 mg/24 h for 1 week. The dose can be increased weekly during Up-Titration Period until either the optimal or the maximal dose of 3 mg/24 h has been reached. Subjects will maintain the optimal/maximal dose during the 2-week Maintenance Period. Following the Maintenance Period, subjects will be de-escalated from their optimal dose by decreasing the dose by 1 mg/24 h every other day during Taper Period until complete withdrawal.
  Other Names: Neupro
  Arms: Rotigotine
Drug: Placebo — Transdermal patch; Patches matching to active treatment patches in size and appearance.
  Up to 3 weeks of Titration,
  2 weeks of Maintenance,
  Up to 4 days of Taper Period.
  Arms: Placebo

SUMMARY:
This is a sleep laboratory study to evaluate the efficacy and safety of Rotigotine in subjects with Restless Legs Syndrome and End-Stage Renal Disease requiring hemodialysis.

The objectives are to demonstrate superiority of Rotigotine against Placebo as well as to investigate the effect of Rotigotine on quality of life and sleep.

ELIGIBILITY:
Inclusion Criteria:

* End-Stage Renal Disease (ESRD) requiring hemodialysis and regular dialysis schedule
* Fulfillment of pre-defined criteria of hematology parameters
* Diagnosis of Restless Legs (RLS) based on the 4 cardinal diagnostic clinical features according to the International Restless Legs Syndrome Study Group
* Initial response to previous dopaminergic treatment for RLS, or has had no previous dopaminergic treatment (ie, de novo)
* Score of ≥ 15 points on the IRLS (indicating moderate to severe RLS) at Baseline
* Score of ≥ 11 points on the RLS-DI (Diagnostic Index) at Baseline
* Score of ≥ 4 points on the Clinical Global Impressions (CGI) Item 1 assessment (indicating moderately ill) at Baseline
* Scores ≥ 15 Periodic Limb Movements (PLMs) per hour on the Periodic Limb Movement Index (PLMI) based on Polysomnography (PSG) (recorded during the second night) as assessed by the investigator at Baseline

Exclusion Criteria:

* Clinically relevant Polyneuropathy or Varicosis which cannot be clearly differentiated from RLS symptoms in the opinion of the investigator
* Clinically relevant concomitant diseases, such as Attention Deficit Hyperactivity Disorder, Painful Legs, and Moving Toes
* Other central nervous system diseases
* Evidence of an impulse control disorder according to the modified Minnesota Impulsive Disorders Interview (mMIDI)
* Lifetime history of suicide attempt (including an active attempt, interrupted attempt, or aborted attempt), or has suicidal ideation in the past 6 months as indicated by a positive response ('yes') to either Question 4 or Question 5 of the Columbia-Suicidality Severity Rating Scale (C-SSRS) at Screening (Visit 1) or Baseline (Visit 2)
* Prior history of psychotic episodes
* History of symptomatic (not asymptomatic) Orthostatic Hypotension
* Clinically relevant Cardiovascular Disease
* Clinically relevant Venous or Arterial Peripheral Vascular Disease
* Malignant Neoplastic Disease requiring therapy within 12 months prior to Screening (Visit 1)
* Treatment with any of the following drug classes: neuroleptics, norepinephrine and dopamine reuptake inhibitors (bupropion), gabapentin, budipine, dopamine antagonist antiemetics (except domperidone), opioids, monoamine oxidase (MAO) inhibitors, catechol-O-methyltransferase (COMT) inhibitors, or psychostimulants (eg, amphetamines)
* Subject is pregnant, nursing, or is a woman of childbearing potential who is not surgically sterile, 2 years postmenopausal, or does not consistently use 2 combined effective methods of contraception (including at least 1 barrier method), unless sexually abstinent
* Previous treatment with dopamine agonists within a period of 14 days prior to Baseline (Visit 2), or L-dopa within 7 days prior to Baseline (Visit 2)
* Medical history indicating intolerability to dopaminergic therapy (if pretreated) or has experienced Augmentation (Garcia-Borreguero and Williams, 2010) when previously treated with any dopaminergic agent
* Subject has received previous treatment with Rotigotine
* Known hypersensitivity to any of the components of the study medication, such as a history of significant Skin Hypersensitivity to adhesives, known Hypersensitivity to other transdermal medications, or unresolved Contact Dermatitis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (15):
- United States (6):
  - 606, Brandon, Florida
  - 604, Newton, Massachusetts
  - 603, West Seneca, New York
  - 607, Dublin, Ohio
  - 605, West Chester, Pennsylvania
  - 601, Austin, Texas
- 101, Innsbruck, Austria
- Finland (2):
  - 201, Helsinki
  - 203, Tampere
- France (2):
  - 302, Bordeaux
  - 301, Montpellier Cédex 5
- Germany (3):
  - 404, Berlin
  - 401, Marburg
  - 402, Schwerin
- 502, Pisa, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment for the SP0934 study began in April 2012. It concluded in October 2013. This was a multicenter study with subjects enrolled by 9 sites across Europe and 6 sites across the United States.
Pre-assignment Details: The participant flow consists of the Randomized Set (RS), which is all subjects randomized into SP0934.
Groups:
- Placebo: Transdermal patch matched according to patch size and appearance.
  Placebo: Transdermal patch; Patches matching to active treatment patches in size and appearance.
  Up to 3 weeks of Titration,
  2 weeks of Maintenance,
  Up to 4 days of Taper Period.
- Rotigotine: Rotigotine Transdermal Patch
  1 mg/24 h, 2 mg/24 h or 3 mg/24 h once daily depending on optimal dose; maximal dose is 3 mg/24 h.
  Subjects start with a Rotigotine dose of 1 mg/24 h for 1 week. The dose can be increased weekly during Up-Titration Period until either the optimal or the maximal dose of 3 mg/24 h has been reached. Subjects will maintain the optimal/maximal dose during the 2-week Maintenance Period. Following the Maintenance Period, subjects will be de-escalated from their optimal dose by decreasing the dose by 1 mg/24 h every other day during Taper Period until complete withdrawal.
Period: Overall Study
Arm/Group | Placebo | Rotigotine
Started | 10 | 20
Completed | 10 | 15
Not Completed | 0 | 5
Not completed — Adverse Event | 0 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population consisted of the Safety Set (SS), which is all subjects who were randomized and had at least 1 patch applied during the Treatment Period.
Groups:
- Placebo: Transdermal patch matched according to patch size and appearance.
  Placebo: Transdermal patch; Patches matching to active treatment patches in size and appearance.
- Total: Total of all reporting groups
Arm/Group | Placebo | Rotigotine | Total
Number analyzed (Participants) | 10 | 20 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (16.3) | 57.2 (12.6) | 55.0 (14.0)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 15 | 23
  >=65 years | 2 | 5 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 7 | 13 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 6 | 8
  White | 4 | 13 | 17
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 5 | 16 | 21
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 6 | 12 | 18
  Europe | 4 | 8 | 12
Weight [Mean (Standard Deviation); unit: Kilograms] | 85.38 (20.99) | 89.42 (15.34) | 88.07 (17.17)
Height [Mean (Standard Deviation); unit: Centimeters] | 171.77 (8.59) | 171.50 (11.99) | 171.59 (10.82)
BMI [Mean (Standard Deviation); unit: kg/ m^2] | 28.850 (6.182) | 30.405 (4.262) | 29.887 (4.931)

OUTCOME MEASURES:

1. Primary Outcome: Ratio From Baseline to the End of the 2-week Maintenance Period in Periodic Limb Movement Index (PLMI)
Description: The PLMI is defined as Periodic Limb Movements (PLMs)/ total time in bed in hours. PLMs are measured by Polysomnography (PSG).
  The reduction of the PLMI is reflected in terms of the ratio from Baseline to the end of the Maintenance Period and was calculated as [PLMI at end of Maintenance Period (MP)] / [PLMI at Baseline].
  A PLMI Ratio <1 indicates an improvement from Baseline to the end of the 2-week MP.
Time Frame: From Baseline over the Up-Titration Period (up to 3 Weeks) to the end of the 2-Week Maintenance Period
Population: Full Analysis Set (FAS), which included all randomized subjects with at least 1 patch applied during the Treatment Period, and had evaluable PSG data at Baseline and at the end of the 2-week Maintenance Period.
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 10 | 15
ratio | 1.16 [0.68 to 1.99] | 0.51 [0.33 to 0.80]
Statistical Analysis 1: Comparison: Placebo vs Rotigotine; Test type: Superiority or Other; p = 0.0232, ANCOVA; An analysis of covariance (ANCOVA) was performed for the log-transformed PLMI ratio with treatment and region as factors and Baseline as a covariate; Treatment Ratio = 0.44, 95% CI 2-sided [0.22 to 0.88]

2. Secondary Outcome: Change From Baseline in the Periodic Limb Movements Index (PLMI) to the End of the Maintenance Period
Description: The PLMI is defined as Periodic Limb Movements (PLMs)/ total time in bed in hours. PLMs are measured by Polysomnography (PSG). A negative value in change from Baseline indicates an improvement from Baseline to the end of the Maintenance Period.
Time Frame: From Baseline over the Up-Titration Period (up to 3 Weeks) to the end of the 2-Week Maintenance Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: movement/ hour
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 10 | 15
movement/ hour | 10.3 (21) | -23.7 (38.7)

3. Secondary Outcome: Change From Baseline in the International Restless Legs Syndrome Study Group Rating Scale (IRLS) Sum Score to the End of the Maintenance Period
Description: The IRLS is a subject based scale that consists of 10 items to evaluate the severity of major RLS symptoms and the impact of the disease on subjects' functioning in daytime activities. Each of the 10 items is measured on a scale that ranges from 0 (not present) to 4 (severe). A sum score between 0 (no RLS symptoms present at all) and 40 (maximum severity in all symptoms) across all 10 items will be calculated.
  A negative value in Change from Baseline indicates an improvement from Baseline in IRLS.
Time Frame: From Baseline over the Up-Titration Period (up to 3 Weeks) to the end of the 2-Week Maintenance Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 10 | 15
units on a scale | -8.6 (7.2) | -15.9 (9.1)

4. Secondary Outcome: Change From Baseline in Clinical Global Impressions (CGI) Item 1 Score
Description: The CGI Item 1 score measures the severity of illness on a scale that ranges from 0 (Not assessed) to 7 (Among the most extremely ill).
Time Frame: Visit 2 (Baseline); Visit 6 (End of Maintence Period)
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Placebo (Visit 2); Placebo (Visit 6): Transdermal patch matched according to patch size and appearance.
  Placebo: Transdermal patch; Patches matching to active treatment patches in size and appearance.
- Rotigotine (Visit 2); Rotigotine (Visit 6): Rotigotine Transdermal Patch
  1 mg/24 h, 2 mg/24 h or 3 mg/24 h once daily depending on optimal dose; maximal dose is 3 mg/24 h.
Arm/Group | Placebo (Visit 2) | Rotigotine (Visit 2) | Placebo (Visit 6) | Rotigotine (Visit 6)
Number analyzed (Participants) | 10 | 15 | 10 | 15
participants
  Not assessed | 0 | 0 | 0 | 0
  Normal, not ill at all | 0 | 0 | 1 | 5
  Borderline ill | 0 | 0 | 1 | 4
  Mildly ill | 0 | 0 | 3 | 3
  Moderately ill | 3 | 3 | 5 | 1
  Markedly ill | 5 | 9 | 0 | 2
  Severely ill | 2 | 2 | 0 | 0
  Among the most extremely ill subjects | 0 | 1 | 0 | 0

5. Secondary Outcome: Change From Baseline in the Restless Legs-6 (RLS-6) Rating Scale 1 to the End of the Maintenance Period
Description: The RLS-6 consists of six scales of which four scales are designed to assess severity of RLS and two scales cover sleep and daytime tiredness.
  Scale 1 measures satisfaction with sleep during the last seven nights on an 11-point scale that ranges between 0 (completely satisfied) to 10 (completely dissatisfied). The ratings are given by the subjects.
  A negative value in Change from Baseline indicates an improvement from Baseline.
Time Frame: From Baseline over the Up-Titration Period (up to 3 Weeks) to the end of the 2-Week Maintenance Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 10 | 15
units on a scale | -1.1 (3.5) | -2.8 (3.2)

6. Secondary Outcome: Change From Baseline in the Restless Legs-6 (RLS-6) Rating Scale 2 to the End of the Maintenance Period
Description: The RLS-6 consists of six scales of which four scales are designed to assess severity of RLS and two scales cover sleep and daytime tiredness.
  Scale 2 measures the severity of RLS symptoms during the last 7 nights in the situation of falling asleep. This is measured on an 11-point scale that ranges between 0 (none) to 10 (very severe). The ratings are given by the subjects.
  A negative value in Change from Baseline indicates an improvement from Baseline.
Time Frame: From Baseline over the Up-Titration Period (up to 3 Weeks) to the end of the 2-Week Maintenance Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 10 | 15
units on a scale | -2.8 (2.9) | -4.4 (2.9)

7. Secondary Outcome: Change From Baseline in the Restless Legs-6 (RLS-6) Rating Scale 3 to the End of the Maintenance Period
Description: The RLS-6 consists of six scales of which four scales are designed to assess severity of RLS and two scales cover sleep and daytime tiredness.
  Scale 3 measures the severity of RLS symptoms during the last seven nights on an 11-point scale that ranges between 0 (none) to 10 (very severe). The ratings are given by the subjects.
  A negative value in Change from Baseline indicates an improvement from Baseline.
Time Frame: From Baseline over the Up-Titration Period (up to 3 Weeks) to the end of the 2-Week Maintenance Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 10 | 15
units on a scale | -3.2 (2.6) | -4.7 (3.1)

8. Secondary Outcome: Change From Baseline in the Restless Legs-6 (RLS-6) Rating Scale 4 to the End of the Maintenance Period
Description: The RLS-6 consists of six scales of which four scales are designed to assess severity of RLS and two scales cover sleep and daytime tiredness.
  Scale 4 measures the severity of RLS symptoms during the last seven days at rest on an 11-point scale that ranges between 0 (none) to 10 (very severe). The ratings are given by the subjects.
  A negative value in Change from Baseline indicates an improvement from Baseline.
Time Frame: From Baseline over the Up-Titration Period (up to 3 Weeks) to the end of the 2-Week Maintenance Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 10 | 15
units on a scale | -1.6 (3.2) | -2.6 (2.2)

9. Secondary Outcome: Change From Baseline in the Restless Legs-6 (RLS-6) Rating Scale 5 to the End of the Maintenance Period
Description: The RLS-6 consists of six scales of which four scales are designed to assess severity of RLS and two scales cover sleep and daytime tiredness.
  Scale 5 measures the severity of RLS symptoms during the last seven days engaged in activities on an 11-point scale that ranges between 0 (none) to 10 (very severe). The ratings are given by the subjects.
  A negative value in Change from Baseline indicates an improvement from Baseline.
Time Frame: From Baseline over the Up-Titration Period (up to 3 Weeks) to the end of the 2-Week Maintenance Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 10 | 15
units on a scale | -1.6 (2.1) | -1.6 (2.7)

10. Secondary Outcome: Change From Baseline in the Restless Legs-6 (RLS-6) Rating Scale 6 to the End of the Maintenance Period
Description: The RLS-6 consists of six scales of which four scales are designed to assess severity of RLS and two scales cover sleep and daytime tiredness.
  Scale 6 measures the severity of daytime tiredness/ sleepiness on an 11-point scale that ranges between 0 (not at all) to 10 (very severe). The ratings are given by the subjects.
  A negative value in Change from Baseline indicates an improvement from Baseline.
Time Frame: From Baseline over the Up-Titration Period (up to 3 Weeks) to the end of the 2-Week Maintenance Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 10 | 15
units on a scale | -1.6 (2.0) | -3.4 (2.3)

11. Secondary Outcome: Change From Baseline in the Periodic Limb Movement During Sleep Arousal Index (PLMSAI) to the End of the Maintenance Period
Description: The Periodic Limb Movement during Sleep Arousal Index (PLMSAI) reflects the influence of the PLM on subject's sleep. Arousal is defined as sudden change in the Electroencephalogram (EEG) activity and the index illustrates to what degree the PLMs contribute to arousal from sleep.
  A negative value in Change from Baseline indicates an improvement from Baseline.
Time Frame: From Baseline over the Up-Titration Period (up to 3 Weeks) to the end of the 2-Week Maintenance Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: movement per hour
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 10 | 15
movement per hour | 4.634 (7.162) | -1.609 (14.412)

12. Secondary Outcome: Change From Baseline in Sleep Efficiency to the End of the Maintenance Period
Description: Sleep stages and time spent in each sleep stage are determined from Electroencephalogram (EEG) readings. Sleep stage data will be used to calculate sleep efficiency. Sleep efficiency will be presented as percentages. Sleep efficiency is the percentage of time in bed spent asleep.
  A postive value in Change from Baseline indicates an improvement from Baseline.
Time Frame: From Baseline over the Up-Titration Period (up to 3 Weeks) to the end of the 2-Week Maintenance Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: sleep time/ total time in bed
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 10 | 15
sleep time/ total time in bed | -2.850 (10.347) | 7.668 (12.317)

13. Secondary Outcome: Change From Baseline in the Restless Legs-Quality of Life (RLS-QoL) Total Score to the End of the Maintenance Period
Description: The RLS-QoL is a disease-specific questionnaire to evaluate quality of life. It consists of 12 items. A total score will be calculated from all of the 12 items. The overall sum score can be from 0 (highest QoL) to 60 (lowest QoL).
  A negative value in Change from Baseline indicates an improvement from Baseline.
Time Frame: From Baseline over the Up-Titration Period (up to 3 Weeks) to the end of the 2-Week Maintenance Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 9 | 15
scores on a scale | -10.2 (10.8) | -10.7 (10.9)

14. Secondary Outcome: Change From Baseline in the Short-Form-36 (SF-36) Item Questionnaire Mental Component Summary (MCS) to the End of the Maintenance Period
Description: The SF-36 is a 36 item generic human research quality of life instrument that uses a recall period of 4 weeks. Items are grouped into 8 domains as follows: Physical Functioning (10 items), Role Physical (4 items), Bodily Pain (2 items), General Health (5 items), Vitality (4 items), Social Functioning (2 items), Role Emotional (3 items), Mental Health (5 items), and a further unscaled single item (question 2) for perceived stability or change in health (Health Transition) during the last year. The norm based scores (based on the US general population) were used for analysis. For the MCS, the lowest and highest possible scores are -9 and 82 (rounded).
  The SF-36 domains (subscores) are scored so that a higher score indicates a better health state.
Time Frame: From Baseline over the Up-Titration Period (up to 3 Weeks) to the end of the 2-Week Maintenance Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 9 | 14
units on a scale | 6.4 (6.6) | 2.2 (10.1)

15. Secondary Outcome: Change From Baseline in the Short-Form-36 (SF-36) Item Questionnaire Physical Component Summary (PCS) to the End of the Maintenance Period
Description: The SF-36 is a 36 item generic human research quality of life instrument that uses a recall period of 4 weeks. Items are grouped into 8 domains as follows: Physical Functioning (10 items), Role Physical (4 items), Bodily Pain (2 items), General Health (5 items), Vitality (4 items), Social Functioning (2 items), Role Emotional (3 items), Mental Health (5 items), and a further unscaled single item (question 2) for perceived stability or change in health (Health Transition) during the last year. The norm-based scores (based on the US general population) were used for analysis. For the PCS, the lowest and highest possible scores are 1 and 81 (rounded).
  The SF-36 domains (subscores) are scored so that a higher score indicates a better health state.
Time Frame: From Baseline over the Up-Titration Period (up to 3 Weeks) to the end of the 2-Week Maintenance Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 9 | 14
units on a scale | -0.3 (8.7) | 3.8 (6.3)

ADVERSE EVENTS:
Time Frame: Adverse Events were recorded during the course of the SP0934 study, which began in April 2012 and concluded in October 2013.
Description: Adverse Events reporting refers to the Safety Set (SS). All subjects who are randomized and have at least 1 patch applied during the Treatment Period were included in the SS.
Arm/Group | Placebo | Rotigotine
Serious Adverse Events (participants affected / at risk) | 1/10 | 3/20
Other Adverse Events (participants affected / at risk) | 4/10 | 12/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Rotigotine (N=20)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Chest pain (General disorders) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Rotigotine (N=20)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Application site pruritus (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Dialysis device complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Electrocardiogram PR prolongation (Investigations) | 0 (0) | 1 (1)
Electrocardiogram ST segment abnormal (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Dysphoria (Psychiatric disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that the results shall be published regardless of outcome.